CLINICAL TRIAL: NCT04930172
Title: A Physician-initiated, National, Multicentre, Ambispective, Observational Registry of Patients Undergoing Branched Endovascular Aortic Procedures With a Total Transfemoral Approach. (TORCH2 Registry)
Brief Title: TOtal tRansfemoral branCHed endovasCular tHoracoabdominal Aortic Repair Registry
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Bertoglio Luca, MD, IRCCS San Raffaele
Other Study IDs: TORCH2
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracic
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Steerable introducers
  Interventions: Device: Steerable introducers

INTERVENTIONS:
Device: Steerable introducers — endografts via total transfemoral approach for visceral vessels cannulation

SUMMARY:
The purpose of the registry is to evaluate the peri-operative, short-, and mid- outcomes of endovascular treatment of thoracoabdominal aneurysms with multibranched endografts via total transfemoral approach for visceral vessels cannulation using steerable sheaths

ELIGIBILITY:
Inclusion Criteria:

* patient adult ( ≥18 years) of either sex,
* patients who underwent a complex aortic procedure requiring a branched endograft via total transfemoral approach in the centers involved in the TORCH2 Registry

Exclusion Criteria:

* patients who did not receive treatment via total transfemoral approach,
* patient with bleeding diathesis or coagulopathy,
* patients with active systemic or cutaneous infection or inflammation,
* patients who are pregnant or lactating,
* patient younger than 18 years of age.
* Absence of at least one imaging follow-up within the first post-operative year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Registry will include approximately 100 patients treated with BEVAR from January 2018 to January 2022 for thoracoabdominal aortic aneurysms with total transfemoral procedures
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
technical success | 30 days
  successful bridging stent graft deployment of all vessels, with aneurysm exclusion, without any signs of type I or type III endoleak, and with no evidence of stenosis/occlusion and mating stent dislocation/kinking at intraoperative completion angiography.
branch instability | 30 days
  freedom from any branch related complications and/or required reinterventions
clinical success | 30 days
  absence of death, type I/III endoleak, graft infection/thrombosis, aneurysm expansion and/or rupture, conversion to open repair, or new treatment-related thoracoabdominal pathologies

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Policlinico S. Orsola Malpighi, Bologna
  - Azienda Universitaria Giuliano Isontina, Cattinara
  - Ospedale Policlinico San Martino, Genova
  - Azienda Ospedaliera di Perugia, Perugia
  - Ospedale San Camillo-Forlanini, Roma
  - Ospedale San Giovanni Addolorata, Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mirza AK, Tenorio ER, Karkkainen JM, Hofer J, Macedo T, Cha S, Ozbek P, Oderich GS. Learning curve of fenestrated and branched endovascular aortic repair for pararenal and thoracoabdominal aneurysms. J Vasc Surg. 2020 Aug;72(2):423-434.e1. doi: 10.1016/j.jvs.2019.09.046. Epub 2020 Feb 17. PMID 32081482
- [Background] Tenorio ER, Oderich GS, Farber MA, Schneider DB, Timaran CH, Schanzer A, Beck AW, Motta F, Sweet MP; U.S. Fenestrated and Branched Aortic Research Consortium Investigators. Outcomes of endovascular repair of chronic postdissection compared with degenerative thoracoabdominal aortic aneurysms using fenestrated-branched stent grafts. J Vasc Surg. 2020 Sep;72(3):822-836.e9. doi: 10.1016/j.jvs.2019.10.091. Epub 2019 Dec 25. PMID 31882309
- [Background] Oikonomou K, Kopp R, Katsargyris A, Pfister K, Verhoeven EL, Kasprzak P. Outcomes of fenestrated/branched endografting in post-dissection thoracoabdominal aortic aneurysms. Eur J Vasc Endovasc Surg. 2014 Dec;48(6):641-8. doi: 10.1016/j.ejvs.2014.07.005. Epub 2014 Aug 28. PMID 25176618
- [Background] Motta F, Parodi FE, Knowles M, Crowner JR, Pascarella L, McGinigle KL, Marston WA, Kibbe MR, Ohana E, Farber MA. Performance of Viabahn balloon-expandable stent compared with self-expandable covered stents for branched endovascular aortic repair. J Vasc Surg. 2021 Feb;73(2):410-416.e2. doi: 10.1016/j.jvs.2020.05.028. Epub 2020 May 27. PMID 32473341
- [Derived] Mario D, Alessandro G, Giovanni P, Gianbattista P, Rocco G, Mauro G, Nicola M, Roberto C, Sandro L, Luca B; TORCH2 Collaborative Study Group. Total Transfemoral Branched Endovascular Thoracoabdominal Aortic Repair (TORCH2): Short-term and 1-Year Outcomes From a National Multicenter Registry. J Endovasc Ther. 2025 Apr;32(2):513-523. doi: 10.1177/15266028231179864. Epub 2023 Jun 16. PMID 37326371